CLINICAL TRIAL: NCT00735839
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Immunogenicity of a Single Dose of Merck S. Aureus Vaccine (V710) in Healthy Male Japanese Subjects
Brief Title: V710 Clinical Study in Healthy Male Japanese Subjects (V710-006) (COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V710-006; 2008_017
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Results first posted 2012-06-26 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Staphylococcal Infection
MeSH Terms: conditions — Staphylococcal Infections | interventions — V710 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- V710 (Experimental): V710 vaccination (60 mcg) single dose on Day 1
  Interventions: Biological: V710
- Placebo (Placebo Comparator): Placebo single dose on Day 1
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: V710 — V710 vaccination (60 mcg, 0.5 ml) single injection on Day 1
  Arms: V710
Biological: Placebo — Saline placebo (0.5 ml) single injection on Day 1
  Arms: Placebo

SUMMARY:
This study is to evaluate the safety and immunogenicity of V710 in Japanese male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Generally Good Physical Health

Exclusion Criteria:

* Received V710 Vaccine, Any Other Investigational S. Aureus Vaccine, Or Investigational S. Aureus Antibodies Before
* Temperature Of Equal/Greater Than 100.4 Degrees F(38 Degrees C) Within The Past 48 Hours

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | V710 | Placebo
Started | 30 | 10
Completed | 30 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V710 | Placebo | Total
Number analyzed (Participants) | 30 | 10 | 40
Age, Customized [Number; unit: participants]
  <20 years | 0 | 0 | 0
  20-74 years | 30 | 10 | 40
  >74 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 30 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Fold Rise (GMFR) From Baseline in Antibody Level
Description: Geometric mean fold rise is calculated as the natural logarithm of the ratio of Day 14 and baseline antibody titers.
Time Frame: Baseline (Day 1) to Day 14 postvaccination
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V710 | Placebo
Number analyzed (Participants) | 30 | 10
Ratio | 4.4 [3.0 to 6.4] | 0.9 [0.8 to 1.0]

2. Primary Outcome: Number of Participants With Vaccine-related Serious Adverse Experiences
Description: Vaccine-related adverse experiences are those determined by the investigator to be possibly, probably, or definitely vaccine-related.
Time Frame: Baseline (Day 1) to Day 84 postvaccination
Measure: Number; unit: Participants
Arm/Group | V710 | Placebo
Number analyzed (Participants) | 30 | 10
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 through Day 14 postvaccination
Arm/Group | V710 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/10
Other Adverse Events (participants affected / at risk) | 12/30 | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V710 (N=30) | Placebo (N=10)
Injection site erythema (General disorders) | 1 (1) | 1 (1)
Injection site pain (General disorders) | 11 (11) | 0 (0)
Injection site swelling (General disorders) | 2 (2) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No